CLINICAL TRIAL: NCT00746824
Title: TM30339: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel, Repeated Subcutaneous Dose-range Study Designed to Determine the Weight Loss in Obese Subjects.
Brief Title: A Study to Determine the Effects of TM30339 on Weight Loss in Obese Individuals.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The IND was withdrawn.
Sponsor: 7TM Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022
Record Dates: First submitted 2008-08-27; First posted 2008-09-04 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Obesity
Keywords: Obesity; weight loss; 7TM Pharma; TM30339; Y4 receptor antagonist
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): AM dose: 0.85 mg
  PM dose: placebo
  Interventions: Drug: TM30339 and/or placebo
- 2 (Experimental): AM dose: 0.85 mg
  PM dose: 0.85 mg
  Interventions: Drug: TM30339 and/or placebo
- 3 (Experimental): AM dose: 2.55 mg
  PM dose: placebo
  Interventions: Drug: TM30339 and/or placebo
- 4 (Experimental): AM dose: placebo
  PM dose: 2.55 mg
  Interventions: Drug: TM30339 and/or placebo
- 5 (Experimental): AM dose: 2.55 mg
  PM dose: 2.55 mg
  Interventions: Drug: TM30339 and/or placebo
- 6 (Experimental): AM dose: placebo
  PM dose: placebo
  Interventions: Drug: TM30339 and/or placebo

INTERVENTIONS:
Drug: TM30339 and/or placebo — The drug and/or placebo will be injected in the abdominal area (site to vary for each injection). Injections will be administered twice daily for 28 days.
  Other Names: 30339

SUMMARY:
The purpose of this study is to determine the effects of TM30339 on weight loss in obese individuals after 28 days dosing.

DETAILED DESCRIPTION:
Obesity is a disease with large socioeconomic consequences and many serious health consequences including Type 2 diabetes, dyslipidemia and cardiovascular diseases. The prevalence of obesity is increasing both in developed and developing countries. There is a great need for further medicinal treatments that effectively will support life style changes or surgical procedures in reducing or maintaining bodyweight.

7TM Pharma has identified TM30339 as a clinical development candidate molecule with potential to assist in the control and amelioration of obesity in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Obese males and females with a BMI of 30-40 kg/m2 inclusive and weight in the range of 85 - 135 kg inclusive
2. Age 18-60 years inclusive
3. Stable lifestyle e.g. smoking, exercise and eating patterns and times for at least 6 months, and willing to maintain these habits during the course of the study
4. Stable weight over past 2 months i.e. a change in body weight < 3 kg as reported by the subject

Exclusion Criteria:

1. Subjects with a history of allergies toward products containing natural rubber (e.g. latex)
2. Subjects with, or with a history of, any clinically significant neurological, gastrointestinal (including bariatric surgery), renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological, or other major disorders
3. Subjects who have a supine blood pressure at screening or Visit 1 higher than 150/95 mmHg by repeat measurements within 15 minutes
4. Subjects who have a QTc (Bazett's correction) interval of > 450 msec at screening
5. Subjects with bradycardia (heart rate < 50)
6. Subjects with heart block
7. Clinically significant thyroid dysfunction as evidenced by TSH > 1.5 X ULN

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change in body weight from baseline (Visit 1) to Visit 5 (the 29th day),which will be computed for each patient and then averaged for each dose arm. | Visit 5 (the 29th day)

SECONDARY OUTCOMES:
To determine the effects of TM30339 after 28 days dosing of obese individuals on: Waist, hip, and waist/hip ratio | Visit 5 (the 29th day)
To determine the effects of TM30339 after 28 days dosing of obese individuals on fasting glucose and insulin, and insulin sensitivity index | Visit 5 (the 29th day)
To determine the effects of TM30339 after 28 days dosing of obese individuals on formation of antibodies towards the drug, TM30339 | Visit 5 (the 29th day)
To determine the effects of TM30339 after 28 days dosing of obese individuals on safety and tolerability | Visit 5 (the 29th day)

REFERENCES:
- See also: 7TM Pharma website — http://www.7tm.com